CLINICAL TRIAL: NCT02476292
Title: Impact of Vasculitis on Employment and Income. An Online Survey of Participants in the VCRC Patient Contact Registry
Brief Title: Impact of Vasculitis on Employment and Income
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: University of Western Ontario, Canada (Other); University of Pennsylvania (Other); University of Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: VCRC 5536
Record Dates: First submitted 2015-06-12; First posted 2015-06-19 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Vasculitis; Systemic Vasculitis; Behcet's Disease; CNS Vasculitis; Cryoglobulinemic Vasculitis; Eosinophilic Granulomatosis; Temporal Arteritis; Wegener Granulomatosis; Henoch-Schoenlein Purpura; Microscopic Polyangiitis; Polyarteritis Nodosa (PAN); Takayasu's Arteritis; Urticarial Vasculitis
MeSH Terms: conditions — Vasculitis; Systemic Vasculitis; Behcet Syndrome; Vasculitis, Central Nervous System; Cryoglobulinemia, Familial Mixed; Giant Cell Arteritis; Granulomatosis with Polyangiitis; IgA Vasculitis; Microscopic Polyangiitis; Polyarteritis Nodosa; Takayasu Arteritis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: online questionnaire — The online questionnaire includes questions about vasculitis, employment and work status before diagnosis and over the course of the disease, work capacity and the financial impact of vasculitis.

SUMMARY:
The purpose of this study is to learn about the impact of vasculitis on employment and income in patients with different systemic vasculitides. All patients enrolled in the Vasculitis Clinical Research Consortium (VCRC) Patient Contact Registry, living in USA or Canada, and followed for more than 1 year since the vasculitis diagnosis will be invited via email to participate in this study, based on an online survey.

DETAILED DESCRIPTION:
All individuals with vasculitis participating in the VCRC contact patient registry, living in the USA or Canada, and with a follow-up period of ≥1 year since the diagnosis of vasculitis will be invited by email to complete an online questionnaire. They will be asked several questions about their disease, their employment and work status before diagnosis and over the course of their disease, their work capacity and the financial impact on their lives.

The survey data will be stored by the Rare Diseases Clinical Research Network's Data Management and Coordinating Center (DMCC) at the University of South Florida. The data will be de-identified. Names or other personal health information will not be collected. If a participant is enrolled in the Vasculitis Patient-Powered Research Network (V-PPRN) University of South Florida (USF) Institutional Review Board Pro00018514, the participant can choose to provide their email address. Upon conclusion of the study period, the data will be sent to the VCRC Principal Investigator and the Protocol 5536 Co-Principal Investigators. All data collected will be sent to the database of Genotypes and Phenotypes (dbGaP) to be stored indefinitely per the Rare Disease Clinical Research Network (RDCRN) Data Sharing Policy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a systemic vasculitis: VCRC Patient Contact Registry includes patients with Behcet's disease, CNS vasculitis, Cryoglobulinemic vasculitis (Cryoglobulinemia), eosinophilic granulomatosis with polyangiitis (Churg-Strauss) (CSS), giant cell (temporal) arteritis (GCA), granulomatosis with polyangiitis (Wegener's) (GPA), Henoch-Schönlein purpura (IgA vasculitis), microscopic polyangiitis (MPA), polyarteritis nodosa (PAN), Takayasu arteritis (TAK), and urticarial vasculitis.
* Age ≥18 years old
* Living in USA or Canada
* Vasculitis diagnosis made ≥1 year ago
* Language requirements: questionnaire will be in English only

Exclusion Criteria:

* Inability to provide informed consent and complete survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals with vasculitis participating in the VCRC Patient Contact Registry, living in the USA or Canada, and with a follow-up period ≥1 year since the diagnosis of vasculitis.
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Percentages of patients with different types of vasculitis who report negative impact of the disease on employment status, productivity, and income. | one day
  Self-reported change in employment status, productivity, and income from the time of diagnosis to the present.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Pagnoux, MD, MPH, MSc, Study Chair — University of Toronto; Peter A. Merkel, MD, MPH, Study Chair — University of Pennsylvania; Lillian Barra, MD, PhD, Study Chair — University of Western Ontario, Canada
Locations (1):
- University of South Florida Data Management and Coordinating Center, Tampa, Florida, United States